CLINICAL TRIAL: NCT05275205
Title: A Phase 2, Prospective, Multicenter, Randomized, Double-Masked, Active-Controlled Study to Assess the Safety, Tolerability, and Evidence of Activity of a Repeat Intravitreal Injection of UBX1325 in Patients With Neovascular Age-Related Macular Degeneration (Wet AMD)
Brief Title: Safety, Tolerability, and Efficacy Study of UBX1325 in Patients With Neovascular Age-Related Macular Degeneration (ENVISION)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UBX1325-03
Record Dates: First submitted 2022-02-17; First posted 2022-03-11 (Actual); Results first posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2023-10

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: Wet AMD
MeSH Terms: interventions — aflibercept; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This study is double-masked, masking patients and investigators to treatment assignment. In addition to this, any Clinical Research Organization and Sponsor team members who are actively engaged with the site will be masked.
  The injector will be unmasked. Some additional roles at the site, Clinical Research Organization and Sponsor levels are unmasked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- UBX1325 (Experimental)
  Interventions: Drug: UBX1325 injection 50 μL
- Aflibercept (EYLEA ®) (Active Comparator)
  Interventions: Drug: EYLEA® (aflibercept) Injection 2 mg (0.05mL)

INTERVENTIONS:
Drug: UBX1325 injection 50 μL — Patients randomized to the UBX1325 arm will receive UBX1325 on Day 1, Weeks 4, 24, and 28
  Arms: UBX1325
Drug: EYLEA® (aflibercept) Injection 2 mg (0.05mL) — Patients randomized to the active-control aflibercept arm will receive aflibercept per label every 8 weeks starting from day 1 until Week 40. In addition, these patients will receive UBX1325 on Week 24 and Week 32; and a sham procedure at Week 4 and Week 28.
  Arms: Aflibercept (EYLEA ®)

SUMMARY:
This study is intended to assess safety, tolerability and biological activity of a repeat IVT injection of UBX1325 in patients with wet AMD.

DETAILED DESCRIPTION:
This is a Phase 2 study. During Screening, every patient will receive a run-in injection of aflibercept. On Day 1, patients will be randomized to either the UBX1325 arm or the aflibercept arm. Patients randomized to the UBX1325 arm will receive UBX1325 on Day 1, Weeks 4, 24, and 28; and sham procedure on Weeks 8, 16, 24, 32, and 40. Patients randomized to the active-control aflibercept arm will receive aflibercept per label every 8 weeks starting from day 1 until Week 40. In addition, these patients will receive UBX1325 on Week 24 and Week 32; and a sham procedure at Week 4 and Week 28.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥50 years.
* Active CNV associated with age-related macular degeneration as evidenced on FA and SD-OCT with presence of intraretinal or subretinal fluid at Screening and Day 1
* BCVA in the study eye (most affected) of 70 to 20 ETDRS letters (equivalent to 20/40 to 20/400 on the Snellen chart) at Screening.
* Patients who have the capacity to give informed consent and who are willing and able to comply with all study-related procedures and assessments.

Exclusion Criteria:

* Concurrent disease in the study eye or structural damage, other than wet AMD, that could compromise BCVA, prevent BCVA improvement, require medical or surgical intervention during the study period, confound interpretation of the results, or interfere with assessment of toxicity or CFP in the study eye.
* Any ocular/intraocular/periocular infection or inflammation in either eye in the past 12 weeks prior to screening
* Subretinal hemorrhage with bleeding area of 4 or greater disc area in the study eye
* History of vitreous hemorrhage in the study eye within 2 months prior to Screening
* Any condition, including laboratory findings and findings in the medical history or in the pre-study assessments, that, in the opinion of the Investigator, constitutes a risk or contraindication for participation in the study or that could interfere with the study objectives, conduct, or evaluation or prevent the patient from fully participating in all aspects of the study
* Significant media opacities, including cataract, which might interfere with VA, assessment of toxicity, or fundus imaging

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Klier, MD, MPH, Study Director — Unity Biotechnology, Inc.
Locations (14):
- United States (14):
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Salehi Retina Institute, Huntington Beach, California
  - Advanced Vision Research Institute, Longmont, Colorado
  - Rand Eye Institute, Deerfield Beach, Florida
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - University Retina and Macula Associates, Lemont, Illinois
  - Illinois Eye Center, Peoria, Illinois
  - Midwest Eye, Carmel, Indiana
  - Mayo Clinic-Rochester, Rochester, Minnesota
  - Sierra Eye Associates, Reno, Nevada
  - EyeHealth Northwest, Portland, Oregon
  - Retina Research Institution of Texas, Abilene, Texas
  - Valley Retina Institute, McAllen, Texas
  - Austin Retina Associates, Round Rock, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | UBX1325 | Aflibercept (EYLEA ®)
Started | 25 | 26
Completed | 19 | 20
Not Completed | 6 | 6
Not completed — Adverse Event | 1 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Death | 1 | 0
Not completed — Patient unable to attend visits | 1 | 0

BASELINE CHARACTERISTICS:
Population: Overall, there were 51 subjects randomized to the study (n=25 in the UBX1325 arm and n=26 in the Aflibercept arm), of which 50 were treated (n=25 in the UBX1325 arm and n=25 in the Aflibercept arm) and which make up the population utilized in specific analyses. Subject 235-3007 was randomized to the Aflibercept arm but did not receive any study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | UBX1325 | Aflibercept (EYLEA ®) | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.3 (8.83) | 78.4 (7.47) | 78.9 (8.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 12 | 13 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 24 | 22 | 46
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 24 | 23 | 47
  Asian | 1 | 1 | 2
  Not reported | 0 | 1 | 1
Study eye [Count of Participants; unit: Participants]
  Left eye (OS) | 16 | 12 | 28
  Right eye (OD) | 9 | 13 | 22
Eye colour [Count of Participants; unit: Participants]
  Blue | 11 | 13 | 24
  Brown | 6 | 9 | 15
  Green | 3 | 0 | 3
  Hazel | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Treatment Emergent Adverse Events (TEAEs) Will be Evaluated for Ocular and Systemic Safety and Tolerability of a Repeat IVT Injection of UBX1325 Compared to Active Control
Description: Ocular and systemic safety and tolerability of a repeat IVT injection of UBX1325 compared to active-control (aflibercept) evaluated by treatment emergent adverse events (TEAEs) through Week 24
Time Frame: Through 24 weeks
Population: The Safety Analysis Set will include all patients who received study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- UBX-1325: UBX1325 injection 50 μL: Patients randomized to the UBX1325 arm will receive UBX1325 on Day 1, Weeks 4, 24, and 28.
- EYLEA® (Aflibercept): EYLEA® (aflibercept) Injection 2 mg (0.05mL): Patients randomized to the active-control aflibercept arm will receive aflibercept per label every 8 weeks starting from day 1 until Week 40. In addition, these patients will receive UBX1325 on Week 24 and Week 32; and a sham procedure at Week 4 and Week 28.
Arm/Group | UBX-1325 | EYLEA® (Aflibercept)
Number analyzed (Participants) | 25 | 25
Participants
  Subjects with At Least One TEAE | 19 | 18
  Cardiac disorders-Atrial fibrillation | 2 | 0
  Cardiac disorders-Angina unstable | 1 | 0
  Cardiac disorders-Cardiac failure congestive | 0 | 1
  Cardiac disorders-Coronary artery disease | 1 | 0
  Endocrine disorders-Hypothyroidism | 1 | 0
  Eye disorders-Neovascular age-related macular degeneration | 5 | 3
  Eye disorders-Conjunctival haemorrhage | 1 | 5
  Eye disorders-Retinal haemorrhage | 4 | 2
  Eye disorders-Macular oedema | 5 | 0
  Eye disorders-Dry eye | 1 | 1
  Eye disorders-Punctate keratitis | 1 | 1
  Eye disorders-Blepharitis | 0 | 1
  Eye disorders-Macular degeneration | 0 | 2
  Eye disorders-Macular thickening | 1 | 0
  Eye disorders-Blindness unilateral | 1 | 0
  Eye disorders-Cataract | 0 | 1
  Eye disorders-Cataract cortical | 0 | 1
  Eye disorders-Diabetic retinopathy | 1 | 0
  Eye disorders-Lacrimation increased | 1 | 0
  Eye disorders-Macular detachment | 1 | 0
  Eye disorders-Optic nerve sheath haemorrhage | 0 | 1
  Eye disorders-Pinguecula | 0 | 1
  Eye disorders-Retinal exudates | 0 | 1
  Eye disorders-Visual acuity reduced | 1 | 0
  Eye disorders-Vitreous haemorrhage | 0 | 1
  Gastrointestinal disorders-Gastrooesophageal reflux disease | 0 | 1
  Gastrointestinal disorders-Hiatus hernia | 1 | 0
  Gastrointestinal disorders-Large intestine polyp | 1 | 0
  Gastrointestinal disorders-Nausea | 1 | 0
  Gastrointestinal disorders-Retroperitoneal haemorrhage | 1 | 0
  Gastrointestinal disorders-Toothache | 0 | 1
  General disorders and administration site conditions-Asthenia | 0 | 1
  General disorders and administration site conditions-Influenza like illness | 0 | 1
  General disorders and administration site conditions-Multiple organ dysfunction syndrome | 1 | 0
  General disorders and administration site conditions-Oedema peripheral | 0 | 1
  Infections and infestations-COVID-19 | 1 | 0
  Infections and infestations-Fungal infection | 0 | 1
  Infections and infestations-Urinary tract infection | 1 | 0
  Injury, poisoning and procedural complications-Corneal abrasion | 1 | 0
  Injury, poisoning and procedural complications-Facial bones fracture | 1 | 0
  Injury, poisoning and procedural complications-Fall | 1 | 0
  Injury, poisoning and procedural complications-Radius fracture | 1 | 0
  Metabolism and nutrition disorders-Dehydration | 1 | 1
  Metabolism and nutrition disorders-Hypoglycaemia | 1 | 0
  Metabolism and nutrition disorders-Hypokalaemia | 0 | 1
  Musculoskeletal and connective tissue disorders-Arthritis | 1 | 0
  Neoplasms benign, malignant and unspecified (incl cysts and polyps)-Meningioma | 0 | 1
  Neoplasms benign, malignant and unspecified (incl cysts and polyps)-Rectal cancer stage III | 1 | 0
  Neoplasms benign, malignant and unspecified (incl cysts and polyps)-Squamous cell carcinoma | 1 | 0
  Nervous system disorders-Carotid arteriosclerosis | 0 | 1
  Renal and urinary disorders-Acute kidney injury | 1 | 0
  Renal and urinary disorders-Renal haematoma | 1 | 0
  Respiratory, thoracic and mediastinal disorders-Chronic obstructive pulmonary -disease | 1 | 0
  Respiratory, thoracic and mediastinal disorders-Rhinitis allergic | 0 | 1
  Surgical and medical procedures-Finger amputation | 0 | 1

2. Secondary Outcome: Change in Best Corrected Visual Acuity (BCVA) From Baseline Over Time
Description: BCVA was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) chart starting at 4 meters.
Time Frame: Through 48 weeks
Population: MMRM Model for BCVA Change from Baseline (Hypothetical Strategy) Full Analysis Set. The hypothetical strategy included all subjects but excluded measurements post anti-VEGF rescue from the analysis.
  The Full Analysis Set included all randomized patients who received study treatment, had a baseline and at least one post baseline BCVA assessment.
Measure: Least Squares Mean (Standard Error); unit: ETDRS Letters
Arm/Group | UBX1325 | Aflibercept (EYLEA ®)
Number analyzed (Participants) | 25 | 25
ETDRS Letters
  Baseline | 58 (13.47) | 62.4 (9.46)
  Week 2: number analyzed (Participants) | 22 | 24
  Week 2 | -0.2 (1.99) | 3.1 (0.85)
  Week 4: number analyzed (Participants) | 24 | 25
  Week 4 | 1.7 (1.45) | 3.0 (1.08)
  Week 8: number analyzed (Participants) | 22 | 25
  Week 8 | 0.6 (1.36) | 3.2 (1.12)
  Week 12: number analyzed (Participants) | 21 | 25
  Week 12 | 1.1 (1.37) | 2.7 (1.5)
  Week 16: number analyzed (Participants) | 13 | 25
  Week 16 | -1.9 (2.87) | 2.2 (1.49)
  Week 20: number analyzed (Participants) | 11 | 25
  Week 20 | 0.7 (1.96) | 2.5 (1.69)
  Week 24: number analyzed (Participants) | 12 | 24
  Week 24 | 0.1 (2.25) | 2.2 (1.42)
  Week 28: number analyzed (Participants) | 11 | 22
  Week 28 | -0.5 (1.86) | 3.2 (1.56)
  Week 32: number analyzed (Participants) | 11 | 21
  Week 32 | -2.4 (1.99) | 2.1 (1.53)
  Week 36: number analyzed (Participants) | 10 | 19
  Week 36 | -4.1 (2.91) | 2.5 (1.43)
  Week 40: number analyzed (Participants) | 9 | 18
  Week 40 | -4.9 (2.38) | 3.4 (1.44)
  Week 44: number analyzed (Participants) | 8 | 19
  Week 44 | -0.5 (2.71) | 1.8 (1.63)
  Week 48: number analyzed (Participants) | 8 | 18
  Week 48 | -1.5 (3.24) | 1.7 (1.73)

3. Secondary Outcome: Change in Central Subfield Thickness (CST) From Baseline Over Time as Assessed by Spectral Domain Optical Coherence Tomography (SD-OCT) and Read by a Central Reading Center
Description: Central Subfield Thickness (CST) measured in microns using spectral domain optical coherence tomography (SD-OCT).
Time Frame: Through 48 weeks
Population: MMRM Model for CST Change from Baseline (Hypothetical Strategy) Full Analysis Set. The hypothetical strategy included all subjects but excluded measurements post anti-VEGF rescue from the analysis.
  The Full Analysis Set included all randomized patients who received study treatment, had a baseline and at least one post baseline BCVA assessment.
Measure: Least Squares Mean (Standard Error); unit: Microns
Arm/Group | UBX1325 | Aflibercept (EYLEA ®)
Number analyzed (Participants) | 25 | 25
Microns
  Baseline | 374.1 (105.72) | 367.5 (151.75)
  Week 2: number analyzed (Participants) | 21 | 24
  Week 2 | 29.9 (10.77) | -35.0 (6.50)
  Week 4: number analyzed (Participants) | 24 | 25
  Week 4 | 56.6 (25.51) | -14.9 (5.89)
  Week 8: number analyzed (Participants) | 22 | 25
  Week 8 | 92.0 (20.52) | 15.2 (8.55)
  Week 12: number analyzed (Participants) | 21 | 25
  Week 12 | 119.6 (25.07) | -18.0 (8.72)
  Week 16: number analyzed (Participants) | 13 | 25
  Week 16 | 85.6 (16.74) | 22.2 (10.14)
  Week 20: number analyzed (Participants) | 11 | 24
  Week 20 | 64.9 (14.74) | -16.4 (7.82)
  Week 24: number analyzed (Participants) | 12 | 23
  Week 24 | 71.2 (13.65) | 31.7 (9.57)
  Week 28: number analyzed (Participants) | 11 | 20
  Week 28 | 94.3 (20.72) | -6.4 (8.33)
  Week 32: number analyzed (Participants) | 10 | 20
  Week 32 | 102.3 (23.61) | 26.4 (9.72)
  Week 36: number analyzed (Participants) | 10 | 19
  Week 36 | 67.8 (16.19) | -29.4 (17.29)
  Week 40: number analyzed (Participants) | 9 | 18
  Week 40 | 66.9 (20.43) | 23.3 (10.77)
  Week 44: number analyzed (Participants) | 8 | 19
  Week 44 | 66.1 (15.23) | -23.3 (7.77)
  Week 48: number analyzed (Participants) | 8 | 18
  Week 48 | 77.2 (16.38) | 28.2 (10.25)

4. Secondary Outcome: Adverse Events (Safety)
Description: Safety is evaluated by incidence of Treatment Emergent Adverse Events (TEAEs).
Time Frame: Through 48 weeks
Population: The Safety Analysis Set will include all patients who received study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | UBX1325 | Aflibercept (EYLEA ®)
Number analyzed (Participants) | 25 | 25
Participants
  Subjects with At Least One TEAE | 20 | 20
  Blood and lymphatic system disorders-Anaemia | 0 | 2
  Cardiac disorders-Atrial fibrillation | 2 | 1
  Cardiac disorders-Angina unstable | 1 | 0
  Cardiac disorders-Arrhythmia supraventricular | 0 | 1
  Cardiac disorders-Cardiac failure congestive | 0 | 1
  Cardiac disorders-Coronary artery disease | 1 | 0
  Cardiac disorders-Ventricular extrasystoles | 0 | 1
  Congenital, familial and genetic disorders-Hydrocele | 0 | 1
  Ear and labyrinth disorders-Vertigo | 1 | 0
  Endocrine disorders-Hypothyroidism | 2 | 0
  Eye disorders-Neovascular age-related macular degeneration | 7 | 7
  Eye disorders-Conjunctival haemorrhage | 1 | 8
  Eye disorders-Retinal haemorrhage | 6 | 3
  Eye disorders-Macular oedema | 5 | 0
  Eye disorders-Macular thickening | 2 | 0
  Eye disorders-Dry eye | 1 | 1
  Eye disorders-Punctate keratitis | 1 | 2
  Eye disorders-Subretinal fluid | 3 | 1
  Eye disorders-Visual acuity reduced | 3 | 1
  Eye disorders-Blepharitis | 0 | 1
  Eye disorders-Cataract | 1 | 1
  Eye disorders-Lacrimation increased | 1 | 0
  Eye disorders-Macular degeneration | 0 | 2
  Eye disorders-Optic nerve sheath haemorrhage | 0 | 2
  Eye disorders-Retinal exudates | 1 | 1
  Eye disorders-Retinal oedema | 2 | 0
  Eye disorders-Vitreous haemorrhage | 0 | 1
  Eye disorders-Blindness unilateral | 1 | 0
  Eye disorders-Cataract cortical | 0 | 1
  Eye disorders-Diabetic retinopathy | 1 | 0
  Eye disorders-Macular detachment | 1 | 0
  Eye disorders-Pinguecula | 0 | 1
  Eye disorders-Posterior capsule opacification | 0 | 1
  Uveitis | 0 | 1
  Visual impairment | 1 | 0
  Gastrointestinal disorders-Nausea | 2 | 2
  Gastrointestinal disorders-Constipation | 0 | 2
  Gastrointestinal disorders-Gastrooesophageal reflux disease | 0 | 2
  Gastrointestinal disorders-Dyspepsia | 0 | 1
  Gastrointestinal disorders-Gingival recession | 0 | 1
  Gastrointestinal disorders-Hiatus hernia | 1 | 0
  Gastrointestinal disorders-Large intestine polyp | 1 | 0
  Gastrointestinal disorders-Retroperitoneal haemorrhage | 1 | 0
  Gastrointestinal disorders-Toothache | 0 | 1
  Gastrointestinal disorders-Vomiting | 1 | 0
  General disorders and administration site conditions-Oedema peripheral | 0 | 2
  General disorders and administration site conditions-Asthenia | 0 | 1
  General disorders and administration site conditions-Influenza like illness | 0 | 1
  General disorders and administration site conditions-Multiple organ dysfunction syndrome | 1 | 0
  General disorders and administration site conditions-Pain | 0 | 1
  Infections and infestations-Urinary tract infection | 1 | 2
  Infections and infestations-COVID-19 | 1 | 2
  Infections and infestations-Nasopharyngitis | 0 | 1
  Infections and infestations-Bacteraemia | 1 | 0
  Infections and infestations-Fungal infection | 0 | 1
  Infections and infestations-Gastrointestinal bacterial infection | 1 | 0
  Infections and infestations-Paronychia | 0 | 1
  Infections and infestations-Pneumonia | 0 | 1
  Infections and infestations-Urosepsis | 0 | 1
  Infections and infestations-Viral rhinitis | 0 | 1
  Injury, poisoning and procedural complications-Fall | 1 | 1
  Injury, poisoning and procedural complications-Skin laceration | 1 | 1
  Injury, poisoning and procedural complications-Corneal abrasion | 1 | 0
  Injury, poisoning and procedural complications-Crush injury | 0 | 1
  Injury, poisoning and procedural complications-Facial bones fracture | 1 | 0
  Injury, poisoning and procedural complications-Femur fracture | 0 | 1
  Injury, poisoning and procedural complications-Fibula fracture | 0 | 1
  Injury, poisoning and procedural complications-Radius fracture | 1 | 0
  Injury, poisoning and procedural complications-Rib fracture | 0 | 1
  Injury, poisoning and procedural complications-Scapula fracture | 0 | 1
  Injury, poisoning and procedural complications-Thoracic vertebral fracture | 0 | 1
  Injury, poisoning and procedural complications-Wrist fracture | 0 | 1
  Investigations-Heart rate irregular | 1 | 1
  Investigations-Electrocardiogram QRS complex abnormal | 1 | 0
  Investigations-QRS axis abnormal | 0 | 1
  Metabolism and nutrition disorders-Dehydration | 1 | 1
  Metabolism and nutrition disorders-Hypokalaemia | 0 | 2
  Metabolism and nutrition disorders-Hyperlipidaemia | 1 | 0
  Metabolism and nutrition disorders-Hypoglycaemia | 1 | 0
  Metabolism and nutrition disorders-Hypomagnesaemia | 0 | 1
  Metabolism and nutrition disorders-Hypovolaemia | 0 | 1
  Musculoskeletal and connective tissue disorders-Arthritis | 1 | 0
  Musculoskeletal and connective tissue disorders-Rhabdomyolysis | 0 | 1
  Neoplasms benign, malignant and unspecified (incl cysts and polyps)-Meningioma | 0 | 1
  Neoplasms benign, malignant and unspecified (incl cysts and polyps)-Rectal cancer stage III | 1 | 0
  Neoplasms benign, malignant and unspecified (incl cysts and polyps)-Squamous cell carcinoma | 1 | 0
  Nervous system disorders-Carotid arteriosclerosis | 0 | 1
  Product issues-Device dislocation | 0 | 1
  Psychiatric disorders-Insomnia | 0 | 1
  Renal and urinary disorders-Acute kidney injury | 1 | 0
  Renal and urinary disorders-Nephropathy | 0 | 1
  Renal and urinary disorders-Renal haematoma | 1 | 0
  Respiratory, thoracic and mediastinal disorders-Asthma | 1 | 0
  Respiratory, thoracic and mediastinal disorders-Chronic obstructive pulmonary disease | 1 | 0
  Respiratory, thoracic and mediastinal disorders-Mediastinal haematoma | 0 | 1
  Respiratory, thoracic and mediastinal disorders-Respiratory failure | 0 | 1
  Respiratory, thoracic and mediastinal disorders-Rhinitis allergic | 0 | 1
  Surgical and medical procedures-Finger amputation | 0 | 1
  Vascular disorders-Hypotension | 1 | 1
  Vascular disorders-Hypertension | 0 | 1

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events by System Organ Class, Preferred Term - Week 0-48 Analysis
Arm/Group | UBX1325 | Aflibercept (EYLEA ®)
All-Cause Mortality (participants affected / at risk) | 1/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 2/25 | 3/25
Other Adverse Events (participants affected / at risk) | 20/25 | 20/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UBX1325 (N=25) | Aflibercept (EYLEA ®) (N=25)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
Crush injury (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Rectal cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Renal haematoma (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | UBX1325 (N=25) | Aflibercept (EYLEA ®) (N=25)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 1
Hypothyroidism (Endocrine disorders) | 2 | 0
Neovascular age-related macular degeneration (Eye disorders) | 7 | 7
Conjunctival haemorrhage (Eye disorders) | 1 | 8
Retinal haemorrhage (Eye disorders) | 6 | 3
Macular oedema (Eye disorders) | 5 | 0
Macular thickening (Eye disorders) | 2 | 0
Punctate keratitis (Eye disorders) | 1 | 2
Subretinal fluid (Eye disorders) | 3 | 1
Visual acuity reduced (Eye disorders) | 3 | 1
Macular degeneration (Eye disorders) | 0 | 2
Optic nerve sheath haemorrhage (Eye disorders) | 0 | 2
Retinal oedema (Eye disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Oedema peripheral (General disorders) | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 2
COVID-19 (Infections and infestations) | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-01-13): https://cdn.clinicaltrials.gov/large-docs/05/NCT05275205/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT05275205/SAP_001.pdf